CLINICAL TRIAL: NCT03456232
Title: High-flux Hemodialysis Versus Hemodiafiltration for End-Stage Renal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDREC2017324H
Record Dates: First submitted 2018-02-27; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Chronic Kidney Failure
Keywords: hemodialysis; hemodiafiltration; end-stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Hemodiafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flux hemodialysis (Experimental): High-flux hemodialysis lasting for 4 hours
  Interventions: Other: High-flux hemodialysis
- Hemodiafiltration (Active Comparator): Hemodiafiltration lasting for 4 hours
  Interventions: Other: Hemodiafiltration

INTERVENTIONS:
Other: High-flux hemodialysis — High-flux hemodialysis using diffusion, ultrafiltration and convection principle to remove harmful substances in the blood and excessive water.
  Arms: High-flux hemodialysis
Other: Hemodiafiltration — Hemodiafiltration is a combination of hemodialysis and hemofiltration with two modes of treatment advantages, both by diffusion and convection principle to remove harmful substances in the blood.
  Arms: Hemodiafiltration

SUMMARY:
This study evaluates the effect of high-flux hemodialysis compared to hemodiafiltration on small and moderate molecule substances clearance. Meanwhile, this study evaluates the effect of high-flux hemodialysis compared to hemodiafiltration on cardiac function. In this self matching study, participants will receive high-flux hemodialysis compared to hemodiafiltration.

DETAILED DESCRIPTION:
Hemodialysis using diffusion, ultrafiltration and convection principle to remove harmful substances in the blood and excessive water, is one of the most commonly replacement therapy.

Hemodiafiltration is a combination of hemodialysis and hemofiltration with two modes of treatment advantages, both by diffusion and convection principle to remove harmful substances in the blood.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has end-stage renal disease.
2. Subject has been on regular dialysis treatment for at least 6 months.
3. Subject has autologous vascular access.
4. Subject is offered thrice weekly hemodialysis.
5. Subject is offered 4 hours duration hemodialysis.

Exclusion Criteria:

1. Infectious disease
2. Poor echocardiographic window that was unsuitable for interpretation

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-03-10 (Estimated); Study Completion 2018-03-20 (Estimated)

PRIMARY OUTCOMES:
Clearance of moderate molecule substance | 4 hours after dialysis
  Clearance rate of b2-microglobulin for one dialysis.

SECONDARY OUTCOMES:
Left ventricular ejection fraction | 4 hours after dialysis
  Left ventricular ejection fraction is calculated by dividing the volume of blood pumped from the left ventricle per beat, also known as stroke volume, by the end-diastolic volume.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi, MD,PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Supporting Information: study protocol, statistic analysis plan, informed consent form, clinical study report.
  Time Frame: Data will be available within 1 year of study completion. Access Criteria: Data access requests will be reviewed by an external Independent Review panel. Requestors will be required to sign a Data Access Agreement.